CLINICAL TRIAL: NCT01224639
Title: Phase I, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Assess the Safety and Immunogenicity of DENVax Vaccine in Healthy Adults
Brief Title: Safety and Immunogenicity Study to Assess TDV, a Live Attenuated Tetravalent Vaccine for Prevention of Dengue Fever
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inviragen Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INV-DEN-102; U1111-1181-8290 (Registry Identifier: WHO)
Record Dates: First submitted 2010-10-09; First posted 2010-10-20 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Dengue Fever
Keywords: dengue fever; live attenuated tetravalent dengue vaccine; TDV; Drug therapy
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: Low Dose; SC (Experimental): TDV-1: 8 x 10^3 Plaque Forming Units (PFU), TDV-2: 5 x 10^3 PFU, TDV-3: 1 x 10^4 PFU, TDV-4: 2 x 10^5 PFU or placebo administered subcutaneously on Days 0 and 90. Dose volume is 0.5 mL.
  Interventions: Biological: TDV - Low Dose
- Group 2: Low Dose; ID (Experimental): TDV-1: 8 x 10^3 PFU, TDV-2: 5 x 10^3 PFU, TDV-3: 1 x 10^4 PFU, TDV-4: 2 x 10^5 PFU or placebo administered intradermally on Days 0 and 90. Dose volume is 0.1 mL.
  Interventions: Biological: TDV - Low Dose
- Group 3: High Dose; SC (Experimental): TDV-1: 2 x 10^4 PFU, TDV-2: 5 x 10^4 PFU, TDV-3: 1 x 10^5 PFU, TDV-4: 3 x 10^5 PFU or placebo administered subcutaneously on Days 0 and 90. Dose volume is 0.5 mL.
  Interventions: Biological: TDV - High Dose
- Group 4: High Dose; ID (Experimental): TDV-1: 2 x 10^4 PFU, TDV-2: 5 x 10^4 PFU, TDV-3: 1 x 10^5 PFU, TDV-4: 3 x 10^5 PFU or placebo administered intradermally on Days 0 and 90. Dose volume is 0.1 mL.
  Interventions: Biological: TDV - High Dose
- Placebo (SC) (Placebo Comparator): Phosphate buffered saline administered subcutaneously in a volume of 0.5 mL.
  Interventions: Biological: Placebo
- Placebo (ID) (Placebo Comparator): Phosphate buffered saline administered intradermally in a dose volume of 0.1 mL.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TDV - Low Dose — TDV is a tetravalent dengue vaccine comprised of four recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. Low dose contains: TDV-1: 8 x 10^3 PFU, TDV-2: 5 x 10^3 PFU, TDV-3: 1 x 10^4 PFU, and TDV-4: 2 x 10^5 PFU, total virus per dose 2.2 x 10^5 PFU
  Other Names: Live attenuated tetravalent dengue vaccine
  Arms: Group 1: Low Dose; SC; Group 2: Low Dose; ID
Biological: TDV - High Dose — TDV is a tetravalent dengue vaccine comprised of four recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. High dose contains TDV-1: 2 x 10^4 PFU, TDV-2: 5 x 10^4 PFU, TDV-3: 1 x 10^5 PFU, and TDV-4: 3 x 10^5 PFU, total virus per dose : 4.7 x 10^5 PFU. TDV administered intradermally.
  Other Names: Live attenuated tetravalent dengue vaccine
  Arms: Group 3: High Dose; SC; Group 4: High Dose; ID
Biological: Placebo — Phosphate Buffered Saline (PBS)
  Other Names: PBS
  Arms: Placebo (ID); Placebo (SC)

SUMMARY:
The purpose of this study is to assess the safety of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) (previously DENVax) in healthy adults when given as either a subcutaneous (SC) or intradermal (ID) injection at two dose levels (low and high). The vaccine will be given as two doses 90 days apart. Safety assessments include injection site evaluation and adverse events. The immune response generated after vaccination will be assessed up to 9 months after the first vaccination.

DETAILED DESCRIPTION:
This is a single center, placebo-controlled, randomized study assessing the safety and tolerability of two dose levels (low and high) of TDV administered subcutaneously or intradermally in two doses separated by an interval of 90 days. Initial dosing of low dose cohort will be performed and Day 21 safety assessed prior to administration of second dose to low dose cohort on Day 90 and initial dosing of high dose cohort. Day 21 safety for the high dose cohort will be assessed prior to administration of second dose for this cohort. Safety (local injection site reactions and solicited and unsolicited adverse events) will be assessed through Day 120 post-first (1 month after the second dose). Immunogenicity will be assessed at specified time points up to Day 120 post-prime (1 month after the second dose) and again on Days 180 and 270 (6 and 9 months post-first).

ELIGIBILITY:
Inclusion Criteria:

* Is male or female aged 18 to 45 years, inclusive, at time of screening.
* Is in good health as determined by medical history, physical examination, and clinical safety laboratory examinations.
* Has body mass index (BMI) in the range 18-27 kilogram per square meter (kg/m^2).
* Has negative serology for Human Immunodeficiency Virus (HIV), Hepatitis C antibody, and Hepatitis B surface antigen.
* Females of child bearing potential must have a negative urine pregnancy test result during screening and a negative urine pregnancy test immediately prior to vaccination and be willing to use oral, implantable, transdermal or injectable contraceptives or another reliable means of contraception approved by the Investigator (intrauterine device, female condom, diaphragm with spermicidal, cervical cap, use of condom by the sexual partner or a sterile sexual partner, or abstinence) from screening until after the last blood sample (at Day 270).
* Is willing and able to give written informed consent to participate.
* Is willing and able to communicate with the Investigator and understand the requirements of the study.

Exclusion Criteria:

* Has any condition which would limit the participant's ability to complete the study.
* Clinically significant hematological, renal, hepatic, pulmonary, central nervous system, cardiovascular or gastrointestinal disorders.
* Has abnormal electrocardiogram (ECG).
* Has febrile illness (temperature greater than or equal to (>=) 38 degree Celsius (°C) or 100.4 degree Fahrenheit (°F) or moderate or severe acute illness or infection within three days of vaccination.
* Diabetes mellitus.
* Has allergy to penicillin, neomycin, streptomycin or gentamicin.
* Hypersensitivity to any vaccine.
* Seropositivity to any of the four dengue serotypes (TDV-1, TDV-2, TDV-3 or TDV-4), yellow fever (YF) virus or West Nile (WN) virus.
* Has previous vaccination (in a clinical trial or with an approved product) against flaviviruses including dengue, YF or WN.
* Has planned vaccination against YF throughout the duration of this study.
* Has receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following each of the vaccinations in this study.
* Travel to dengue-endemic areas in the two months prior to study start or planned travel to dengue-endemic areas during the study period, including low altitude regions of Colombia where dengue is endemic.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months prior to the first vaccination, or long- term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 0.5 milligram per kilogram per day [mg/kg/day]) prior to the first vaccination.
* Has a history of recurring migraines or on prescription medication for treatment of recurring headaches or migraines.
* Use of any non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen or antihistamines for the 3 days immediately prior to each vaccination.
* Use of prescription or over the counter medications 7 days before the first vaccination (Day 0), excluding contraceptives and painkillers containing NSAIDs or acetaminophen, cold remedies, hormone replacement and antihistamines.
* Positive urine screen for cocaine, amphetamines, opiates, or cannabinoids.
* Receipt of any other investigational product or participation in any other clinical trial in the month before the first vaccination (Day 0) or during the conduct of this study.
* Receipt of blood products or immunoglobulins 8 weeks before the first vaccination (Day 0) or planned use during the study period.
* Donation of blood 6 weeks before the first vaccination (Day 0) or at any time during the study.
* Females who are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-10-11 (Actual); Primary Completion 2011-06-09 (Actual); Study Completion 2011-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan D Velez, MD, Ph.D., Principal Investigator — PECET, Universidad the Antioquia, Medellin, Colombia
Locations (1):
- Program For The Study and Control of Tropical Diseases, Medellín, Colombia

REFERENCES:
- [Derived] Osorio JE, Velez ID, Thomson C, Lopez L, Jimenez A, Haller AA, Silengo S, Scott J, Boroughs KL, Stovall JL, Luy BE, Arguello J, Beatty ME, Santangelo J, Gordon GS, Huang CY, Stinchcomb DT. Safety and immunogenicity of a recombinant live attenuated tetravalent dengue vaccine (DENVax) in flavivirus-naive healthy adults in Colombia: a randomised, placebo-controlled, phase 1 study. Lancet Infect Dis. 2014 Sep;14(9):830-8. doi: 10.1016/S1473-3099(14)70811-4. Epub 2014 Jul 23. PMID 25087476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Colombia from 11 October 2010 to 09 November 2011.
Pre-assignment Details: Healthy male and female participants were enrolled in 1 of the 8 treatment groups: Low Dose Subcutaneous:TDV, Low Dose Subcutaneous: Placebo, Low Dose Intradermal:TDV, Low Dose Intradermal:Placebo, High Dose Subcutaneous:TDV, High Dose Subcutaneous:Placebo, High Dose Intradermal:TDV, High Dose Intradermal:Placebo.
Groups:
- Low Dose Subcutaneous: TDV: TDV 0.5 milliliter (mL), injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). Takeda's Tetravalent Dengue Vaccine Candidate (TDV) (previously DENVax) comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. Low dose contains: TDV-1: 8*10^3 plaque forming units (PFU), TDV-2: 5*10^3 PFU, TDV-3: 1*10^4 PFU, and TDV-4: 2*10^5 PFU, total virus per dose: 2.2*10^5 PFU.
- Low Dose Subcutaneous: Placebo; High Dose Subcutaneous: Placebo: TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
- Low Dose Intradermal: TDV: TDV 0.1 mL, injection, intradermally, once on Day 0 (first dose) and Day 90 (second dose). TDV is a tetravalent dengue vaccine comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. Low dose contains: TDV-1: 8*10^3 PFU, TDV-2: 5*10^3 PFU, TDV-3: 1*10^4 PFU, and TDV-4: 2*10^5 PFU, total virus per dose: 2.2*10^5 PFU.
- Low Dose Intradermal: Placebo; High Dose Intradermal: Placebo: TDV placebo-matching 0.1 mL injection, intradermally, once on Day 0 (first dose) and Day 90 (second dose).
- High Dose Subcutaneous: TDV: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV is a tetravalent dengue vaccine comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. High dose contains TDV-1: 2*10^4 PFU, TDV-2: 5*10^4 PFU, TDV-3: 1*10^5 PFU, and TDV-4: 3*10^5 PFU, total virus per dose: 4.7*10^5 PFU.
- High Dose Intradermal: TDV: TDV 0.1 mL, injection, intradermally, once on Day 0 (first dose) and Day 90 (second dose). TDV is a tetravalent dengue vaccine comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. High dose contains TDV-1: 2*10^4 PFU, TDV-2: 5*10^4 PFU, TDV-3: 1*10^5 PFU, and TDV-4: 3*10^5 PFU, total virus per dose: 4.7*10^5 PFU.
Period: Overall Study
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Started | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
Completed | 19 | 5 | 21 | 3 | 19 | 4 | 17 | 3
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received at least one dose of study vaccine and for whom post-dosing safety data was obtained.
Groups:
- Low Dose Subcutaneous: TDV: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV is a tetravalent dengue vaccine comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4. Low dose contains: TDV-1: 8*10^3 PFU, TDV-2: 5*10^3 PFU, TDV-3: 1*10^4 PFU, and TDV-4: 2*10^5 PFU, total virus per dose: 2.2*10^5 PFU.
- Total: Total of all reporting groups
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo | Total
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5 | 96
Age, Customized [Number; unit: participants]
  Less than (<) 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Greater than or equal to (>=) 18 and <65 years | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5 | 96
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 11 | 2 | 17 | 3 | 12 | 4 | 67
  Male | 5 | 1 | 10 | 1 | 4 | 1 | 6 | 1 | 29
Race/Ethnicity, Customized [Number; unit: participants] — The baseline measure category "other" refers to mixed race.
  participants
    White | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 7
    Other | 17 | 5 | 17 | 3 | 21 | 4 | 18 | 4 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Injection Site Reaction by Severity
Description: Solicited local reactions were reported using a participant diary. Pain was categorized as Mild (aware of pain but it does not interfere with daily activity and no pain medication is taken); Moderate (aware of pain; there is interference with daily activity or it requires use of pain medication); Severe (aware of pain and it prevents daily activity), redness was categorized as Mild (greater than [>] 15 millimeter [mm]); Moderate as (15-30 mm); Severe (>30 mm), swelling was categorized as Mild (<15 mm); Moderate (15-30 mm); Severe (>30 mm), and itching was categorized as Mild (slight itching at injection site); Moderate (moderate itching at injection extremity); Severe (itching over entire body).
Time Frame: Within 14 days after either of the vaccination given on Day 1 or 90 (Day 14 for first vaccination, Day 104 for second vaccination)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
participants
  Pain: Mild | 12 | 1 | 8 | 2 | 8 | 0 | 10 | 1
  Pain: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Redness: Mild | 1 | 0 | 12 | 0 | 1 | 1 | 5 | 0
  Redness: Moderate | 1 | 0 | 8 | 0 | 5 | 0 | 9 | 0
  Redness: Severe | 4 | 0 | 0 | 0 | 7 | 0 | 3 | 0
  Swelling: Mild | 0 | 0 | 10 | 0 | 2 | 0 | 5 | 0
  Swelling: Moderate | 2 | 0 | 4 | 0 | 2 | 0 | 5 | 0
  Swelling: Severe | 4 | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Itching: Mild | 4 | 0 | 12 | 1 | 7 | 1 | 13 | 1
  Itching: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Systemic Adverse Events (AEs) by Severity
Description: Solicited systemic AEs were reported using a participant diary. Solicited systemic AEs included fever (>= 37.8°C), headache, muscle pain, joint pain, eye pain, photophobia, fatigue, body rash, nausea, vomiting and other (any other symptom not listed in the diary) and were categorized as Mild: transient symptoms, discomfort noticed but easily tolerated, no interference to normal daily activities; Moderate: marked symptoms, moderate interference with daily activities; Severe: considerable interference with daily activities.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
participants
  Fever: Mild | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0
  Fever: Moderate | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
  Fever: Severe | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Headache: Mild | 4 | 1 | 12 | 2 | 9 | 0 | 6 | 2
  Headache: Moderate | 7 | 1 | 4 | 0 | 2 | 1 | 5 | 1
  Headache: Severe | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Muscle pain: Mild | 10 | 0 | 3 | 2 | 4 | 0 | 6 | 0
  Muscle pain: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Muscle pain: Severe | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Joint pain: Mild | 4 | 0 | 2 | 0 | 3 | 0 | 3 | 0
  Joint pain: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint pain: Severe | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Eye pain: Mild | 6 | 2 | 8 | 1 | 4 | 1 | 7 | 1
  Eye pain: Moderate | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Eye pain: Severe | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Photophobia: Mild | 5 | 1 | 6 | 1 | 2 | 1 | 3 | 2
  Photophobia: Moderate | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Photophobia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue: Mild | 9 | 2 | 7 | 1 | 5 | 0 | 10 | 4
  Fatigue: Moderate | 3 | 0 | 4 | 0 | 2 | 0 | 2 | 0
  Fatigue: Severe | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Body Rash: Mild | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 0
  Body Rash: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Body Rash: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Nausea: Mild | 4 | 2 | 4 | 1 | 4 | 0 | 4 | 2
  Nausea: Moderate | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0
  Nausea: Severe | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  Vomiting: Severe | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Other: Mild | 4 | 0 | 2 | 0 | 6 | 1 | 4 | 1
  Other: Moderate | 2 | 1 | 4 | 0 | 4 | 1 | 2 | 2
  Other: Severe | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Local and Systemic AEs
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
participants
  Local solicited AEs | 15 | 1 | 20 | 2 | 14 | 1 | 18 | 1
  Systemic solicited AEs | 17 | 4 | 17 | 2 | 17 | 3 | 17 | 4

4. Primary Outcome: Number of Participants With Unsolicited Local and Systemic AEs
Time Frame: Baseline up to 30 days after second vaccination (Day 120)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
participants
  Local unsolicited AEs | 0 | 0 | 3 | 0 | 1 | 0 | 4 | 0
  Systemic unsolicited AEs | 18 | 5 | 16 | 3 | 16 | 2 | 14 | 3

5. Secondary Outcome: Geometric Mean Neutralizing Antibody Titers (GMTs) of All Four Dengue Serotypes After First Vaccination
Description: GMT was assessed for the four dengue serotypes: Dengue TDV-1, TDV-2, TDV-3 and TDV-4. GMTs and 95 percent (%) confidence interval (CIs) were calculated by taking the anti-logs of the means and 95% CI of the log transformed titers.
Time Frame: Days 14, 30, 60 and 90 after first vaccination
Population: The full analysis set (FAS) included all randomized participants who received at least one dose of study vaccine and for whom valid pre- and post-dosing blood samples were received. Here 'n' is number of participants with non-missing microneutralization (MN) Assay samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
titer
  Day 14 TDV-1 (n=19, 5, 21, 3, 21, 4, 18, 5) | 12.45 [8.32 to 18.61] | 5.00 [5.00 to 5.00] | 22.08 [12.64 to 38.58] | 5.00 [5.00 to 5.00] | 111.29 [58.46 to 211.83] | 5.00 [5.00 to 5.00] | 72.66 [27.52 to 191.86] | 5.00 [5.00 to 5.00]
  Day 14 TDV-2 (n=19, 5, 21, 3, 21, 4, 18, 5) | 6.94 [4.31 to 11.19] | 5.00 [5.00 to 5.00] | 7.43 [4.89 to 11.29] | 5.00 [5.00 to 5.00] | 6.73 [4.72 to 9.59] | 5.00 [5.00 to 5.00] | 7.64 [3.39 to 17.20] | 5.00 [5.00 to 5.00]
  Day 14 TDV-3 (n=19, 5, 21, 3, 21, 4, 18, 5) | 17.93 [8.20 to 39.17] | 5.00 [5.00 to 5.00] | 20.00 [9.17 to 43.60] | 5.00 [5.00 to 5.00] | 26.04 [12.30 to 55.13] | 5.00 [5.00 to 5.00] | 117.58 [41.32 to 334.54] | 5.00 [5.00 to 5.00]
  Day 14 TDV-4 (n=19, 5, 21, 3, 21, 4, 18, 5) | 7.75 [5.02 to 11.96] | 5.00 [5.00 to 5.00] | 11.04 [6.26 to 19.46] | 5.00 [5.00 to 5.00] | 5.71 [4.72 to 6.90] | 5.00 [5.00 to 5.00] | 11.22 [5.40 to 23.32] | 5.00 [5.00 to 5.00]
  Day 30 TDV-1(n=19, 5, 21, 3, 21, 4, 18, 5) | 49.79 [26.00 to 95.36] | 5.00 [5.00 to 5.00] | 48.76 [27.94 to 85.09] | 5.00 [5.00 to 5.00] | 208.37 [102.74 to 422.61] | 5.00 [5.00 to 5.00] | 153.96 [80.16 to 295.69] | 5.00 [5.00 to 5.00]
  Day 30 TDV-2 (n=19, 5, 21, 3, 21, 4, 18, 5) | 363.60 [73.44 to 1800.07] | 5.00 [5.00 to 5.00] | 475.52 [88.35 to 2559.42] | 5.00 [5.00 to 5.00] | 8682.13 [5174.46 to 14567.58] | 5.00 [5.00 to 5.00] | 2370.24 [718.63 to 7817.74] | 5.00 [5.00 to 5.00]
  Day 30 TDV-3 (n=19, 5, 21, 3, 21, 4, 18, 5) | 25.82 [9.77 to 68.26] | 5.00 [5.00 to 5.00] | 67.83 [25.66 to 179.29] | 5.00 [5.00 to 5.00] | 42.03 [22.35 to 79.05] | 5.00 [5.00 to 5.00] | 307.91 [115.76 to 819.04] | 5.00 [5.00 to 5.00]
  Day 30 TDV-4 (n=19, 5, 21, 3, 21, 4, 18, 5) | 33.33 [14.01 to 79.31] | 5.00 [5.00 to 5.00] | 57.51 [21.68 to 152.57] | 5.00 [5.00 to 5.00] | 9.06 [4.89 to 16.79] | 5.00 [5.00 to 5.00] | 22.88 [10.76 to 48.69] | 5.00 [5.00 to 5.00]
  Day 60 TDV-1 (n=19, 5, 21, 3, 19, 4, 18, 5) | 49.79 [23.98 to 103.39] | 5.00 [5.00 to 5.00] | 38.70 [19.18 to 78.08] | 6.30 [2.33 to 17.02] | 103.28 [50.97 to 209.26] | 5.00 [5.00 to 5.00] | 86.40 [39.48 to 189.10] | 5.00 [5.00 to 5.00]
  Day 60 TDV-2 (n=19, 5, 21, 3, 19, 4, 18, 5) | 230.44 [66.23 to 801.82] | 5.00 [5.00 to 5.00] | 262.51 [63.99 to 1076.87] | 5.00 [5.00 to 5.00] | 1280.00 [768.38 to 2132.27] | 5.00 [5.00 to 5.00] | 838.01 [375.38 to 1870.77] | 5.00 [5.00 to 5.00]
  Day 60 TDV-3 (n=19, 5, 21, 3, 19, 4, 18, 5) | 34.57 [14.13 to 84.59] | 5.00 [5.00 to 5.00] | 50.40 [20.72 to 122.56] | 5.00 [5.00 to 5.00] | 30.99 [18.33 to 52.37] | 5.00 [5.00 to 5.00] | 148.14 [50.82 to 431.83] | 5.00 [5.00 to 5.00]
  Day 60 TDV-4 (n=19, 5, 21, 3, 19, 4, 18, 5) | 13.39 [7.04 to 25.46] | 5.00 [5.00 to 5.00] | 26.48 [10.42 to 67.30] | 5.00 [5.00 to 5.00] | 5.58 [4.43 to 7.02] | 5.00 [5.00 to 5.00] | 10.60 [5.31 to 21.13] | 5.00 [5.00 to 5.00]
  Day 90 TDV-1 (n=19, 5, 21, 3, 19, 4, 17, 3) | 34.57 [16.17 to 73.92] | 5.00 [5.00 to 5.00] | 43.44 [18.91 to 99.80] | 5.00 [5.00 to 5.00] | 109.09 [49.55 to 240.18] | 5.00 [5.00 to 5.00] | 80.00 [33.72 to 189.78] | 5.00 [5.00 to 5.00]
  Day 90 TDV-2 (n=19, 5, 21, 3, 19, 4, 17, 3) | 181.80 [55.42 to 596.40] | 5.00 [5.00 to 5.00] | 309.61 [94.50 to 1014.43] | 5.00 [5.00 to 5.00] | 1912.01 [1254.58 to 2913.94] | 5.00 [5.00 to 5.00] | 666.63 [305.13 to 1456.45] | 5.00 [5.00 to 5.00]
  Day 90 TDV-3 (n=19, 5, 21, 3, 19, 4, 17, 3) | 30.99 [13.75 to 69.81] | 5.00 [5.00 to 5.00] | 60.43 [27.22 to 134.18] | 5.00 [5.00 to 5.00] | 34.57 [20.61 to 57.99] | 5.00 [5.00 to 5.00] | 135.92 [51.41 to 359.33] | 5.00 [5.00 to 5.00]
  Day 90 TDV-4 (n=19, 5, 21, 3, 19, 4, 17, 3) | 11.16 [6.11 to 20.38] | 5.00 [5.00 to 5.00] | 28.29 [11.62 to 68.86] | 5.00 [5.00 to 5.00] | 6.22 [5.12 to 7.56] | 5.00 [5.00 to 5.00] | 11.30 [5.86 to 21.81] | 5.00 [5.00 to 5.00]

6. Secondary Outcome: GMTs of All Four Dengue Serotypes After Second Vaccination
Description: GMT was assessed for the four dengue serotypes: TDV-1, TDV-2, TDV-3 and TDV-4. GMTs and 95% CIs were calculated by taking the anti-logs of the means and 95% CI of the log transformed titers.
Time Frame: Days 14 and 30 after second vaccination (Day 104 and 120 respectively)
Population: The FAS included all randomized participants who received at least one dose of study vaccine and for whom valid pre- and post-dosing blood samples were received. Here 'n' is number of participants with non-missing MN Assay samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
titer
  Day 104 TDV-1 (n=19, 5, 21, 3, 18, 4, 17, 3) | 111.09 [45.46 to 271.46] | 5.00 [5.00 to 5.00] | 137.92 [68.77 to 276.60] | 5.00 [5.00 to 5.00] | 244.39 [133.53 to 447.30] | 5.00 [5.00 to 5.00] | 230.93 [131.23 to 406.38] | 5.00 [5.00 to 5.00]
  Day 104 TDV-2 (n=19, 5, 21, 3, 18, 4, 17, 3) | 222.18 [76.63 to 644.18] | 5.00 [5.00 to 5.00] | 341.84 [102.43 to 1140.85] | 5.00 [5.00 to 5.00] | 1382.48 [935.89 to 2042.17] | 5.00 [5.00 to 5.00] | 589.88 [277.32 to 1254.75] | 5.00 [5.00 to 5.00]
  Day 104 TDV-3 (n=19, 5, 21, 3, 18, 4, 17, 3) | 73.03 [33.64 to 158.56] | 5.00 [5.00 to 5.00] | 144.92 [81.49 to 257.70] | 5.00 [5.00 to 5.00] | 63.50 [45.45 to 88.71] | 5.00 [5.00 to 5.00] | 250.56 [127.21 to 493.50] | 5.00 [5.00 to 5.00]
  Day 104 TDV-4 (n=19, 5, 21, 3, 18, 4, 17, 3) | 21.51 [11.58 to 39.95] | 5.00 [5.00 to 5.00] | 72.46 [35.46 to 148.05] | 5.00 [5.00 to 5.00] | 10.39 [7.09 to 15.24] | 5.00 [5.00 to 5.00] | 27.71 [14.56 to 52.77] | 5.00 [5.00 to 5.00]
  Day 120 TDV-1(n=19, 5, 21, 3, 19, 4, 17, 3) | 128.55 [52.36 to 315.60] | 5.00 [5.00 to 5.00] | 92.81 [47.92 to 179.77] | 5.00 [5.00 to 5.00] | 181.82 [101.33 to 326.24] | 5.00 [5.00 to 5.00] | 160.00 [91.07 to 281.09] | 5.00 [5.00 to 5.00]
  Day 120 TDV-2 (n=19, 5, 21, 3, 19, 4, 17, 3) | 206.55 [64.16 to 664.90] | 5.00 [5.00 to 5.00] | 314.76 [95.01 to 1042.74] | 5.00 [5.00 to 5.00] | 1536.13 [972.63 to 2426.11] | 5.00 [5.00 to 5.00] | 543.69 [248.70 to 1188.55] | 5.00 [5.00 to 5.00]
  Day 120 TDV-3 (n=19, 5, 21, 3, 19, 4, 17, 3) | 69.14 [33.72 to 141.77] | 5.00 [5.00 to 5.00] | 88.33 [46.17 to 168.99] | 5.00 [5.00 to 5.00] | 78.56 [49.89 to 123.70] | 5.00 [5.00 to 5.00] | 271.84 [126.94 to 582.17] | 5.00 [5.00 to 5.00]
  Day 120 TDV-4 (n=19, 5, 21, 3, 19, 4, 17, 3) | 20.74 [10.59 to 40.64] | 5.00 [5.00 to 5.00] | 48.76 [24.58 to 96.74] | 5.00 [5.00 to 5.00] | 9.64 [6.41 to 14.51] | 5.00 [5.00 to 5.00] | 16.99 [9.34 to 30.90] | 5.00 [5.00 to 5.00]

7. Secondary Outcome: Rate of Seroconversion to Each of Four Dengue Serotypes After the First Vaccination
Description: Seroconversion was defined as a Plaque Reduction Neutralization Test (PRNT) titer resulting in 50% reduction in plaques (PRNT[50]) >=10 (if the pre-vaccination PRNT[50] value was <10, indicated as a value of 5 in the immunogenicity data collection sheet) OR a PRNT(50) value that was >=4-fold the pre-vaccination titer value (if the pre-vaccination PRNT[50] value was >=10). Seroconversion was assessed for the four dengue serotypes: TDV-1, TDV-2, TDV-3 and TDV-4. The 95% CIs for percentages are the exact CIs (%) based upon the binomial distribution. Percentages are based on the number of participants in the FAS with non-missing MN assay samples at each visit.
Time Frame: Days 14, 30, 60 and 90 after first vaccination
Population: The FAS included all randomized participants who received at least one dose of study vaccine and for whom valid pre- and post-dosing blood samples were received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
percentage of participants
  Day 14 TDV-1 (n=19, 5, 21, 3, 21, 4, 18, 5) | 63.2 [38.4 to 83.7] | 0 [0.0 to 52.2] | 66.7 [43.0 to 85.4] | 0 [0.0 to 70.8] | 90.5 [69.8 to 98.8] | 0 [0.0 to 60.2] | 83.3 [58.6 to 96.4] | 0 [0.0 to 52.2]
  Day 14 TDV-2 (n=19, 5, 21, 3, 21, 4, 18, 5) | 10.5 [1.3 to 33.1] | 0 [0.0 to 52.2] | 19.0 [5.4 to 41.9] | 0 [0 to 70.8] | 14.3 [3.0 to 36.3] | 0 [0.0 to 60.2] | 11.1 [1.4 to 34.7] | 0 [0.0 to 52.2]
  Day 14 TDV-3 (n=19, 5, 21, 3, 21, 4, 18, 5) | 52.6 [28.9 to 75.6] | 0 [0.0 to 52.2] | 42.9 [21.8 to 66.0] | 0 [0.0 to 70.8] | 52.4 [29.8 to 74.3] | 0 [0.0 to 60.2] | 83.3 [58.6 to 96.4] | 0 [0.0 to 52.2]
  Day 14 TDV-4 (n=19, 5, 21, 3, 21, 4, 18, 5) | 21.1 [6.1 to 45.6] | 0 [0.0 to 52.2] | 33.3 [14.6 to 57.0] | 0 [0.0 to 70.8] | 9.5 [1.2 to 30.4] | 0 [0.0 to 60.2] | 38.9 [17.2 to 64.3] | 0 [0.0 to 52.2]
  Day 30 TDV-1 (n=19, 5, 21, 3, 21, 4, 18, 5) | 89.5 [66.9 to 98.7] | 0 [0.0 to 52.2] | 90.5 [69.6 to 98.8] | 0 [0.0 to 70.8] | 95.2 [76.2 to 99.9] | 0 [0.0 to 60.2] | 100 [81.5 to 100.0] | 0 [0.0 to 52.2]
  Day 30 TDV-2 (n=19, 5, 21, 3, 21, 4, 18, 5) | 68.4 [43.4 to 87.4] | 0 [0.0 to 52.2] | 66.7 [43.0 to 85.4] | 0 [0.0 to 70.8] | 100.0 [83.9 to 100.0] | 0 [0.0 to 60.2] | 88.9 [65.3 to 98.6] | 0 [0.0 to 52.2]
  Day 30 TDV-3 (n=19, 5, 21, 3, 21, 4, 18, 5) | 57.9 [33.5 to 79.7] | 0 [0.0 to 52.2] | 71.4 [47.8 to 88.7] | 0 [0.0 to 70.8] | 81.0 [58.1 to 94.6] | 0 [0.0 to 60.2] | 94.4 [72.7 to 99.9] | 0 [0.0 to 52.2]
  Day 30 TDV-4 (n=19, 5, 21, 3, 21, 4, 18, 5) | 63.2 [38.4 to 83.7] | 0 [0.0 to 52.2] | 71.4 [47.8 to 88.7] | 0 [0.0 to 70.8] | 23.8 [8.2 to 47.2] | 0 [0.0 to 60.2] | 66.7 [41.0 to 86.7] | 0 [0.0 to 52.2]
  Day 60 TDV-1 (n=19, 5, 21, 3, 19, 4, 18, 5) | 89.5 [66.9 to 98.7] | 0 [0.0 to 52.2] | 81.0 [58.1 to 94.6] | 33.3 [0.8 to 90.6] | 94.7 [74.0 to 99.9] | 0 [0.0 to 60.2] | 100 [81.5 to 100.0] | 0 [0.0 to 52.2]
  Day 60 TDV-2 (n=19, 5, 21, 3, 19, 4, 18, 5) | 78.9 [54.4 to 93.6] | 0 [0.0 to 52.2] | 66.7 [43.0 to 85.4] | 0 [0.0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0.0 to 60.2] | 94.4 [72.7 to 99.9] | 0 [0.0 to 52.2]
  Day 60 TDV-3 (n=19, 5, 21, 3, 19, 4, 18, 5) | 63.2 [38.4 to 83.7] | 0 [0.0 to 52.2] | 66.7 [43.0 to 85.4] | 0 [0.0 to 70.8] | 89.5 [66.9 to 98.7] | 0 [0.0 to 60.2] | 88.9 [65.3 to 98.6] | 0 [0.0 to 52.2]
  Day 60 TDV-4 (n=19, 5, 21, 3, 19, 4, 18, 5) | 47.4 [24.4 to 71.1] | 0 [0.0 to 52.2] | 42.9 [21.8 to 66.0] | 0 [0.0 to 70.8] | 5.3 [0.1 to 26.0] | 0 [0.0 to 60.2] | 33.3 [13.3 to 59.0] | 0 [0.0 to 52.2]
  Day 90 TDV-1 (n=19, 5, 21, 3, 19, 4, 17, 3) | 73.7 [48.8 to 90.9] | 0 [0.0 to 52.2] | 71.4 [47.8 to 88.7] | 0 [0.0 to 70.8] | 94.7 [74.0 to 99.9] | 0 [0.0 to 60.2] | 88.2 [63.6 to 98.5] | 0 [0.0 to 70.8]
  Day 90 TDV-2 (n=19, 5, 21, 3, 19, 4, 17, 3) | 73.7 [48.8 to 90.9] | 0 [0.0 to 52.2] | 76.2 [52.8 to 91.8] | 0 [0.0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0.0 to 60.2] | 94.1 [71.3 to 99.9] | 0 [0.0 to 70.8]
  Day 90 TDV-3 (n=19, 5, 21, 3, 19, 4, 17, 3) | 68.4 [43.4 to 87.4] | 0 [0.0 to 52.2] | 76.2 [52.8 to 91.8] | 0 [0.0 to 70.8] | 94.7 [74.0 to 99.9] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 90 TDV-4 (n=19, 5, 21, 3, 19, 4, 17, 3) | 36.8 [16.3 to 61.6] | 0 [0.0 to 52.2] | 52.4 [29.8 to 74.3] | 0 [0.0 to 70.8] | 26.3 [9.1 to 51.2] | 0 [0.0 to 60.2] | 41.2 [18.4 to 67.1] | 0 [0.0 to 70.8]

8. Secondary Outcome: Rate of Seroconversion to Each of Four Dengue Serotypes After the Second Vaccination
Description: Seroconversion was defined as a PRNT titer resulting in 50% reduction in plaques (PRNT[50]) >=10 (if the pre-vaccination PRNT[50] value was <10, indicated as a value of 5 in the immunogenicity data collection sheet) OR a PRNT(50) value that was >=4-fold the pre-vaccination titer value (if the pre-vaccination PRNT[50] value was >=10). Seroconversion was assessed for the four dengue serotypes: TDV-1, TDV-2, TDV-3 and TDV-4. The 95% CIs for percentages are the exact CIs (%) based upon the binomial distribution. Percentages are based on the number of participants in the FAS with non-missing MN assay samples at each visit (n).
Time Frame: Days 14 and 30 after second vaccination (Days 104 and 120 respectively)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
percentage of participants
  Day 104 TDV-1 (n=19, 5, 21, 3, 18, 4, 17, 3) | 89.5 [66.9 to 98.7] | 0 [0.0 to 52.2] | 100.0 [83.9 to 100.0] | 0 [0.0 to 70.8] | 100.0 [81.5 to 100.0] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 104 TDV-2 (n=19, 5, 21, 3, 18, 4, 17, 3) | 78.9 [54.4 to 93.9] | 0 [0.0 to 52.2] | 76.2 [52.8 to 91.8] | 0 [0.0 to 70.8] | 100.0 [81.5 to 100.0] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 104 TDV-3 (n=19, 5, 21, 3, 18, 4, 17, 3) | 84.2 [60.4 to 96.6] | 0 [0.0 to 52.2] | 100.0 [83.9 to 100.0] | 0 [0.0 to 70.8] | 100.0 [81.5 to 100.0] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 104 TDV-4 (n=19, 5, 21, 3, 18, 4, 17, 3) | 73.7 [48.8 to 90.9] | 0 [0.0 to 52.2] | 90.5 [69.6 to 98.8] | 0 [0.0 to 70.8] | 55.6 [30.8 to 78.5] | 0 [0.0 to 60.2] | 88.2 [63.6 to 98.5] | 0 [0.0 to 70.8]
  Day 120 TDV-1 (n=19, 5, 21, 3, 19, 4, 17, 3) | 94.7 [74.0 to 99.9] | 0 [0.0 to 52.2] | 100.0 [83.9 to 100.0] | 0 [0.0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 120 TDV-2 (n=19, 5, 21, 3, 19, 4, 17, 3) | 78.9 [54.4 to 93.6] | 0 [0.0 to 52.2] | 76.2 [52.8 to 91.8] | 0 [0.0 to 70.8] | 100.0 [81.5 to 100.0] | 0 [0.0 to 60.2] | 94.1 [71.3 to 99.9] | 0 [0.0 to 70.8]
  Day 120 TDV-3 (n=19, 5, 21, 3, 19, 4, 17, 3) | 94.7 [74.0 to 99.9] | 0 [0.0 to 52.2] | 95.2 [76.2 to 99.9] | 0 [0.0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 120 TDV-4 (n=19, 5, 21, 3, 19, 4, 17, 3) | 73.7 [48.8 to 90.9] | 0 [0.0 to 52.2] | 95.2 [76.2 to 99.9] | 0 [0.0 to 70.8] | 47.4 [24.4 to 71.1] | 0 [0.0 to 60.2] | 76.5 [50.1 to 93.2] | 0 [0.0 to 70.8]

9. Secondary Outcome: Percentage of Participants With Durability of Immune Response
Description: Immune response was considered durable if the participant had detectable neutralizing antibodies (seroconversion) to all 4 dengue serotypes at 90 and 180 days after the second dose (i.e. Days 180 and 270, respectively). Seroconversion is defined as post-vaccination PRNT(50) titer >=10 where pre-vaccination PRNT 50 titer <10, or post-vaccination PRNT(50) Titer >=4-fold the pre-vaccination PRNT(50) titer value where pre-vaccination PRNT(50) titer >=10. Percentage of participants with seroconversion on Days 180 and 270 are based on the number of participants in the FAS with non-missing MN assay samples at each visit. The 95% CIs for percentages are the exact CIs (%) based upon the binomial distribution.
Time Frame: Days 180 and 270
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 19 | 4 | 17 | 3
percentage of participants
  Day 180 TDV-1 | 78.9 [54.4 to 93.9] | 0 [0 to 52.2] | 90.5 [69.6 to 98.8] | 0 [0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0 to 70.8]
  Day 180 TDV-2 | 73.7 [48.8 to 90.9] | 0 [0.0 to 52.2] | 81.0 [58.1 to 94.6] | 0 [0.0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0.0 to 60.2] | 94.1 [71.3 to 99.9] | 0 [0.0 to 70.8]
  Day 180 TDV-3 | 94.7 [74.0 to 99.9] | 20.0 [0.5 to 71.6] | 100.0 [83.9 to 100.0] | 0 [0.0 to 70.8] | 94.7 [74.0 to 99.9] | 0 [0.0 to 60.2] | 100.0 [80.5 to 100.0] | 0 [0.0 to 70.8]
  Day 180 TDV-4 | 63.2 [38.4 to 83.7] | 0 [0.0 to 52.2] | 71.4 [47.8 to 88.7] | 0 [0.0 to 70.8] | 31.6 [12.6 to 56.6] | 0 [0.0 to 60.2] | 52.9 [27.8 to 77.0] | 0 [0.0 to 70.8]
  Day 270 TDV-1 | 68.4 [43.4 to 87.4] | 0 [0 to 52.2] | 66.7 [43.0 to 85.4] | 0 [0 to 70.8] | 89.5 [66.9 to 98.7] | 0 [0 to 60.2] | 94.1 [71.3 to 99.9] | 0 [0 to 70.8]
  Day 270 TDV-2 | 73.7 [48.8 to 90.9] | 0 [0.0 to 52.2] | 81.0 [58.1 to 94.6] | 0 [0.0 to 70.8] | 100.0 [82.4 to 100.0] | 0 [0.0 to 60.2] | 94.1 [71.3 to 99.9] | 0 [0.0 to 70.8]
  Day 270 TDV-3 | 68.4 [43.4 to 87.4] | 0 [0.0 to 52.2] | 76.2 [52.8 to 91.8] | 0 [0.0 to 70.8] | 57.9 [33.5 to 79.7] | 0 [0.0 to 60.2] | 88.2 [63.6 to 98.5] | 0 [0.0 to 70.8]
  Day 270 TDV-4 | 42.1 [20.3 to 66.5] | 0 [0.0 to 52.2] | 57.1 [34.0 to 78.2] | 0 [0.0 to 70.8] | 15.8 [3.4 to 39.6] | 0 [0.0 to 60.2] | 35.3 [14.2 to 61.7] | 0 [0.0 to 70.8]

10. Secondary Outcome: Number of Participants Positive for Vaccine Viremia for Each of the Four Vaccine Strain Serotypes After the First and Second Vaccination
Description: Serotype-specific vaccine viremia was assessed for the four vaccine strain serotypes: TDV-1, TDV-2, TDV-3 and TDV-4. Only those serotypes and time-points where at least 1 participant had serotype-specific vaccine viremia detection were reported.
Time Frame: Baseline and at multiple time points up to Day 14 after each vaccination
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 19 | 5 | 21 | 3 | 21 | 4 | 18 | 5
participants
  Day 5 TDV-2 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Day 7 TDV-2 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 1 | 0 | 2 | 0 | 6 | 0 | 4 | 0
  Day 9 TDV-2 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 5 | 0 | 6 | 0 | 9 | 0 | 5 | 0
  Day 11 TDV-2 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 4 | 0 | 7 | 0 | 17 | 0 | 5 | 0
  Day 14 TDV-2 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 3 | 0 | 3 | 0 | 10 | 0 | 8 | 0
  Day 97 TDV-2 (n= 19, 5, 21, 3, 21, 3, 17, 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 99 TDV-2 (n= 19, 5, 21, 3, 21, 3, 17, 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 101 TDV-2 (n= 19, 5, 21, 3, 21, 3, 17, 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 104 TDV-2 (n= 19, 5, 21, 3, 18, 4, 17, 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5 TDV-3 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 7 TDV-3 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Day 9 TDV-3 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 97 TDV-3 (n= 19, 5, 21, 3, 19, 4, 17, 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 99 TDV-3 (n= 19, 5, 21, 3, 19, 4, 17, 3) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 101 TDV-3 (n= 19, 5, 21, 3, 19, 4, 17, 3) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 7 TDV-4 (n= 19, 5, 21, 3, 21, 4, 18, 5) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 97 TDV-4 (n= 19, 5, 21, 3, 19, 4, 17, 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Duration of Vaccine Viremia
Time Frame: 14 Days after each vaccination
Population: Due to the low prevalence of vaccine viremia, estimates of average titer duration of viral RNA within study groups would not be meaningful. Therefore as per change in planned analysis only number of participants with positive vaccine viremia of all four vaccine strain serotypes after first and second vaccination was reported.
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Titers of Vaccine Viremia
Time Frame: 14 Days after each vaccination
Population: Due to the low prevalence of vaccine viremia, estimates of average titer levels of viral RNA within study groups would not be meaningful. Therefore as per change in planned analysis only number of participants with positive vaccine viremia of all four vaccine strain serotypes after first and second vaccination was reported.
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are adverse events that started after the first dose of double-blind study vaccine and up to Day 120
Description: A SAE is any untoward medical occurrence that at any dose was fatal, life-threatening, required hospitalization/prolongation of existing hospitalization, resulted in persistent/significant disability/incapacity, congenital anomaly/birth defect, medically significant or required intervention to prevent one or other of the outcomes listed here.
Arm/Group | Low Dose Subcutaneous: TDV | Low Dose Subcutaneous: Placebo | Low Dose Intradermal: TDV | Low Dose Intradermal: Placebo | High Dose Subcutaneous: TDV | High Dose Subcutaneous: Placebo | High Dose Intradermal: TDV | High Dose Intradermal: Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/5 | 0/21 | 1/3 | 1/21 | 0/4 | 0/18 | 0/5
Other Adverse Events (participants affected / at risk) | 12/19 | 5/5 | 13/21 | 3/3 | 15/21 | 2/4 | 13/18 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Subcutaneous: TDV (N=19) | Low Dose Subcutaneous: Placebo (N=5) | Low Dose Intradermal: TDV (N=21) | Low Dose Intradermal: Placebo (N=3) | High Dose Subcutaneous: TDV (N=21) | High Dose Subcutaneous: Placebo (N=4) | High Dose Intradermal: TDV (N=18) | High Dose Intradermal: Placebo (N=5)
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Subcutaneous: TDV (N=19) | Low Dose Subcutaneous: Placebo (N=5) | Low Dose Intradermal: TDV (N=21) | Low Dose Intradermal: Placebo (N=3) | High Dose Subcutaneous: TDV (N=21) | High Dose Subcutaneous: Placebo (N=4) | High Dose Intradermal: TDV (N=18) | High Dose Intradermal: Placebo (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EYE PAIN (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PHOTOPHOBIA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
INJECTION SITE HAEMATOMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PYERXIA (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
VACCINATION SITE HAEMATOMA (General disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 0
VACCINATION SITE SCAB (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 2 | 4 | 0 | 5 | 0 | 4 | 1
ORAL HERPES (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1
VAGINITIS BACTERIAL (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD FIBRINOGEN INCREASED (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 4 | 1 | 6 | 1 | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PERIPHERAL COLDNESS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.